CLINICAL TRIAL: NCT01513772
Title: The Effect of Dexmedetomidine on the Emergence Agitation in Nasal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, So Yeon Kim, Clinical assistant professor, Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 4-2011-0742
Record Dates: First submitted 2012-01-16; First posted 2012-01-20 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Airway Extubation
MeSH Terms: interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Control (Placebo Comparator)
  Interventions: Drug: Normal saline 0.9%
- Dexmedetomidine (Active Comparator)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine(4㎍/mL) : 0.4㎍/kg/hr infusion until extubation
  Arms: Dexmedetomidine
Drug: Normal saline 0.9% — Normal saline(guess as 4㎍/mL) : 0.4㎍/kg/hr infusion until extubation
  Arms: Control

SUMMARY:
The investigators examined the effect of dexmedetomidine on the emergence agitation and postoperative quality of recovery in nasal surgery

DETAILED DESCRIPTION:
Emergence agitation during the immediate postanesthetic period is common. It may lead to serious consequences for the patient, such as injury, increased pain, hemorrhage, self-extubation, and removal of catheters. Emergence agitation is common in ENT surgery. The aim of this study is to evaluate the effect of dexmedetomidine on the emergence agitation and postoperative quality of recovery in adult patients undergoing nasal surgery.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 20,
* ASA class I and II,
* nasal surgery

Exclusion Criteria:

* bradycardia (< 45 bpm),
* heart block,
* liver failure,
* renal failure,
* uncontrolled hypertension,
* body mass index ≥ 30 kg/m2

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2012-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Emergence agitation | 20min

SECONDARY OUTCOMES:
Postoperative quality of recovery | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine and Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea